CLINICAL TRIAL: NCT03835988
Title: Geniculate Artery Embolization for Knee Osteoarthritis
Acronym: GAEKO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid department protocol prevented patient recruitment and affected funding.
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Ani Mirakhur, Clinical Assistant Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB19-0007
Record Dates: First submitted 2019-01-31; First posted 2019-02-11 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Osteo Arthritis Knee
Keywords: Embolization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Geniculate Artery Embolization (Experimental): Patients undergoing geniculate artery embolization. Patients will be assessed and followed post-procedurally to detect changes in knee pain and function. Medication use, adverse events and performance based tests of physical function will also be recorded. A pre-procedural MRI will be compared to a 6 month post-procedure MRI to assess for changes in synovitis and assess for complications.
  Interventions: Device: Geniculate Artery Embolization

INTERVENTIONS:
Device: Geniculate Artery Embolization — Embolization is a procedure completed by an Interventional Radiologist in which abnormal blood vessels are blocked for treatment purposes. In the case of geniculate artery embolization, abnormal blood vessels which supply your knee joint are blocked in an effort to reduce inflammation and subsequently and reduce pain and improve joint function.
  Other Names: Embozene Embolic Particles; Embosphere Embolic Particles

SUMMARY:
A prospective cohort study to study the effectiveness and safety profile of geniculate artery embolization for the treatment of symptomatic knee osteoarthritis.

DETAILED DESCRIPTION:
Purpose: The investigators aim to determine whether geniculate artery embolization is a safe treatment for symptomatic knee osteoarthritis and confirm published reports of sustained post-procedural pain relief, improved physical function and investigate potential improvements in joint function quantitatively through imaging and targeted assessments.

Participants:Twenty patients with moderate to severe knee pain, pain refractory for 3 months of conservative therapies, imaging features of symptomatic osteoarthritis and ineligible for arthroplasty for 1 year.

Procedures (methods): Patients will undergo a brief clinical evaluation to verify eligibility through inclusion and exclusion criteria in addition to a comprehensive joint pain treatment history will be recorded including active analgesic and anti-inflammatory use. A pre-procedural MRI will be completed to assess the extent of their osteoarthritis, signs of active synovitis and vascular anatomy of the knee. Evaluations post geniculate artery embolization will occur at 24 hours, 1, 6 and 12 months to assess for changes in knee pain and joint function and monitor adverse events. An MRI will be performed at the 6 month visit to detect changes in synovitis and exclude complications.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe knee pain (visual analog scale (VAS) > 50 mm), and
* Pain refractory for at least 3 months of conservative therapies (anti-inflammatory drugs, physical therapy, muscle strengthening or intra-articular injections), and
* Kellgren-Lawrence grade 1, 2 or 3 on knee radiograph, and
* MRI features of active synovitis (Synovial thickening and/or enhancement on MRI using pre-gadolinium sagittal T2-weighted/proton-density sequences and post-gadolinium T1 weighted imaging, respectively), and
* Willing, able and mentally competent to provide written informed consent (to ensure that all study subjects demonstrate an understanding of the risks of the procedure and participate in the informed consent), and
* Not eligible for surgical arthroplasty within 1 year of estimated procedure date

Exclusion Criteria:

* Major surgery within the past six weeks (excluding arthroscopic/meniscal interventions), or
* Ipsilateral knee intra-articular injection in the last 3 months, or
* Pregnant or attempting to become pregnant during study period, or
* Current local infection, or
* Life expectancy less than 6 months, or
* Known advanced atherosclerosis, or
* Rheumatoid or seronegative arthropathies, or
* Infectious arthritis, or
* Prior knee surgery (excluding arthroscopic/meniscal interventions), or
* Uncorrectable coagulopathy including international normalized ratio (INR) > 1.5 or platelets < 50,000, or
* Iodinated contrast allergy resulting in anaphylaxis, or
* Inability to lay supine on an angiographic table >500 lbs due to table weight limits, or
* Renal dysfunction as defined as glomerular filtration rate < 30 mL/min/1.73m2 obtained within the past 30 days, or
* Patients with documented noncompliance with previous medical care, or
* Patients with certain psychiatric disorders such as schizophrenia, borderline personality disorder, uncontrolled depression, or mental/cognitive impairment that limits the individual's ability to understand the proposed therapy, or
* Absence of synovitis on MRI

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Pain (mm): visual analog scale | 1 year
  Severity of pain as assessed by visual analog scale. The visual analog scale is a 100 mm horizontal line with 0 mm correlating with "No Pain" and 100 mm with "Worst Possible Pain". Accompanying the verbal description is an illustrative guide correlating values to facial expressions. Patients mark their responses with a single vertical line. Results will be recorded prior to the procedure and afterwards at each follow-up visit to measure for changes in knee pain.
Patient function (arbitrary units) | 1 year
  Knee injury and Osteoarthritis Outcome Score (KOOS) will be used to measure joint function. This is a questionnaire in which questions regarding pain, other symptoms, function in activities of daily living, function in sport and recreation and knee-related quality of life are answered to calculate subscale scores. Each subscale (symptoms, activities of daily living, sport and recreation, quality of life) is scored from 0 to 100 with 0 representing extreme symptoms and 100 indicating no symptoms). The questionnaire will be completed at follow-up evaluations to measure change in each subscale from baseline (prior to intervention). Investigators will analyze scores to determine if patient's subjective joint function changes.

SECONDARY OUTCOMES:
Medication use (arbitrary units) | 1 year
  Change in number or dosage of osteoarthritis medical therapy including oral, topical medications and joint injections will be recorded. Number will be defined as total number of medications used for knee osteoarthritis. Dosage will be defined as the frequency of administration multiplied by the dose of each administration (i.e. 200 mg, 3 times daily will be scored as 600 mg daily). Values will be recorded at each follow-up visit to measure change from baseline and summarized with simple statistics (i.e. percentage of patients with a decrease in medication use).
Physical function (arbitrary units) | 1 year
  Change in physical function performance will be assessed with a 30 second chair stand test.
Synovitis (arbitrary units) | 1 year
  A semiquantifiable synovitis scoring scale on contrast enhanced MRI will be used to assess change in synovitis as proposed by Guermazi et al. in 2011. Synovial thickness will be scored semiquantifiably from grade 0 to 2 at 11 anatomical locations. Grading is calculate by meausrement of maximal synovial thickness with 2 mm or less scored as grade 0, 2-4 mm as grade 1 and > 4 mm as grade 2. Grading at each location are summed to compute a total synovitis score with a minimum score of 0 representing no synovitis and a maximal score of 22 representing severe synovitis. Investigators will compare scores calculated at a 6 month contrast enhanced MRI to those obtained prior to intervention to assess for changes in synovitis.

OTHER OUTCOMES:
Patient complications (arbitrary units) | 1 year
  The number of complications or adverse events with associated descriptions from geniculate artery embolization will be recorded. Results will be summarized using simple statistics.

CONTACTS AND LOCATIONS:
Locations (1):
- South Healthy Campus, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] Guermazi A, Roemer FW, Hayashi D, Crema MD, Niu J, Zhang Y, Marra MD, Katur A, Lynch JA, El-Khoury GY, Baker K, Hughes LB, Nevitt MC, Felson DT. Assessment of synovitis with contrast-enhanced MRI using a whole-joint semiquantitative scoring system in people with, or at high risk of, knee osteoarthritis: the MOST study. Ann Rheum Dis. 2011 May;70(5):805-11. doi: 10.1136/ard.2010.139618. Epub 2010 Dec 27. PMID 21187293